CLINICAL TRIAL: NCT05680324
Title: the Aesthetic and Functional Impact of Monsplasty in Women Undergoing Abdominoplasty
Brief Title: Impact of Monsplasty in Women Undergoing Abdominoplasty
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mostafa Mohamed Hassan, Resident doctor, Assiut University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MMhassan
Record Dates: First submitted 2022-12-26; First posted 2023-01-11 (Actual); Last update posted 2023-01-11 (Actual); Status verified 2022-12

CONDITIONS: Liposuction; Mons Pubis Lift
Keywords: monsplasty

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Abdominoplasty with Monsplasty (Active Comparator)
  Interventions: Procedure: Monsplasty
- Abdominoplasty without monsplasty (Active Comparator)
  Interventions: Procedure: Monsplasty

INTERVENTIONS:
Procedure: Monsplasty — liposuction assisted monsplasty

SUMMARY:
Evaluate The aesthetic and function satisfaction outcomes of different monsplasty surgery with or after abdominoplasty

DETAILED DESCRIPTION:
The high incidence of female obesity has resulted in common complaints of a large mons pubis and labia majora (outer labial lips) related to unsightly fat deposits. The mons and labia majora enlarge, protrude, descend, and hang. Even with dramatic weight loss, these areas remain descended and bulky, with excess fat and skin. The affected majora can cause difficulty with sexual intercourse and maintenance of hygiene, and result in discomfort when wearing pants and swimsuits. These unnatural .fat deposits can also severely affect self-esteem

The surgical treatment of the enlarged mons pubis and labia majora has been poorly understood and therefore often neglected. Traditionally, the mons has been treated by fat reduction, whether by liposuction or open excision, along with a pubic skin lift. However, skin elevation is usually unsatisfactory, because the mons will descend again upon standing. Many of these unsuccessful lifts present after a simultaneous abdominoplasty.

In many ways, the treatment of the mons pubis correlates with the treatment of the hidden penis in the obese or formerly obese male.1-3 Excess suprapubic skin and mons fat removal-along with tacking of the fibrofatty tissue of the pubic skin flap to the rectus fascia-are mandatory to achieve a lasting, successful mons pubis lift.4 Labia majora reduction. Depends on the surgically appropriate removal of fat and/or skin

ELIGIBILITY:
Inclusion Criteria:

* Any adult married woman from 20 to 45 years old candidate for abdominoplasty with stable weight in last 6 months

Exclusion Criteria:

* patients less than 20 years old and more than 45 years old
* patients with medical conditions affecting wound healing
* patients with skin infection in lower abdomen and pubic area

Ages: 20 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 24 (Estimated)
Dates: Start 2021-10-10 (Actual); Primary Completion 2023-04 (Estimated); Study Completion 2023-05 (Estimated)

PRIMARY OUTCOMES:
Determine better result | 3 years
  Determine which is bettereither abdominoplast with monsplasty or abdominoplasty alone by a questionnaire

CONTACTS AND LOCATIONS:
Locations (1):
- Assiut university, Asyut, Egypt